CLINICAL TRIAL: NCT06110988
Title: A Clinical Study for Pan-vascular Interventional Control System in Percutaneous Coronary Intervention
Brief Title: A Clinical Study for the Pan-vascular Interventional Robotic System
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shenzhen Institute of Advanced Biomedical Robot Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Ge Junbo, Chief of Cardiology, Shanghai Zhongshan Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P02-IIT-KSI
Record Dates: First submitted 2023-10-25; First posted 2023-11-01 (Actual); Last update posted 2024-04-26 (Actual); Status verified 2024-04

CONDITIONS: Percutaneous Coronary Intervention; Pan-vascular Interventional Robotic System

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pan-vascular interventional robotic system (Experimental): Pan-vascular interventional robotic system assisted PCI
  Interventions: Device: Pan-vascular interventional robotic system

INTERVENTIONS:
Device: Pan-vascular interventional robotic system — Pan-vascular interventional robotic system assited PCI for delivery and manipulation of guidewires, catheters, and quick exchange balloon dilatation catheters/stents.

SUMMARY:
The goal of this prospective, single-center, single-arm study is to explore the efficacy and safety of the pan-vascular interventional robotic system for percutaneous coronary intervention (PCI), researchers will assess the clinical success, technical success, and record the intraoperative data (PCI time, guidewire operation time, dose of contrast medium, radiation exposure doses, etc). All subjects will be followed up on the day of surgery, before discharge (or 48 hours after surgery) and 1 month after surgery to observe the safety indicators.

ELIGIBILITY:
Inclusion Criteria:

1. General Inclusion criteria:

1. 18 years old ≤ age ≤80 years old;
2. have a clinical indication for PCI (clinical evidence of ischemic heart disease or a positive functional study);
3. Subjects or their legal representative has been informed of the nature of the study, signed informed consent and were willing to cooperate in the follow-up.

2. Angiographic inclusion criteria:

1. study lesion is a single de novo native coronary artery lesion (previously untreated coronary artery disease);
2. target vessel diameter between 2.5 mm and 4.0 mm;
3. single lesion length ≤38 mm, with at least 2.0 mm normal segments on the proximal and distal edges of the lesion;
4. stenosis ≥50% and < 100%.

Exclusion Criteria:

1. General exclusion criteria:

1. hemodynamic instability (including hypotension or use of vasopressors to maintain blood pressure);
2. STEMI, cardiopulmonary resuscitation, or cardiogenic shock within 7 days before surgery;
3. subjects were required to undergo planned PCI or CABG within 30 days after surgery, or had undergone PCI within 72 hours before surgery, or had undergone PCI within 30 days before surgery with a protocol-defined major adverse coronary event (MACE) or serious adverse event (SAE);
4. subjects had a stroke or transient ischemic attack (TIA) within 30 days before surgery;
5. subjects with active peptic ulcer or upper GI bleeding within 6 months before surgery;
6. The study lesion requires planned treatment with directional coronary atherectomy (DCA), laser, rotational atherectomy or any device except for balloon dilatation prior to stent placement
7. left ventricular ejection fraction (LVEF) < 35%;
8. subjects with known allergies to or contraindications to antiplatelet drugs, anticoagulants, stent materials and their coatings, or allergies to contrast agents, unable to receive adequate preoperative medication or manage with clinically appropriate alternatives;
9. subjects had a history of bleeding tendency or coagulopathy or refused blood transfusion;
10. severe liver and kidney dysfunction;
11. patients who are scheduled to undergo additional cardiac surgery (e.g., valve replacement or cardiac ablation) within 30 days after surgery;
12. inaccessible vascular access (radial artery/femoral artery) or severe vascular stenosis, occlusion or skin infection at the puncture site;
13. uncontrolled severe infection;
14. subjects participating in clinical studies of other devices or drugs during the same period;
15. pregnant and lactating women of childbearing age;
16. subjects judged by the investigator to be ineligible for the study.

2. Exclusion criteria for angiography:

1. in-stent restenosis or any previous stent placement within 5.0 mm (proximal or distal) of the target lesion；
2. bifurcation lesions, in which the target vessel branch needs to be protected but cannot be protected;
3. the target lesion is located at the ostium or anastomosis of coronary artery;
4. investigate evidence of intravascular thrombosis;
5. severe tortuosity or calcification of the proximal end of the study vessel or target lesion;
6. study the complete occlusion of the lesion;
7. Target lesion located in left main coronary artery, or unprotected left main coronary artery disease (> 50% stenosis in left main coronary artery).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Estimated)
Dates: Start 2024-04-30 (Estimated); Primary Completion 2024-09-30 (Estimated); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
Clinical Success | Discharge or 48 hours post intervention, whichever comes first
  Less than 30% residual stenosis (visual estimate) post PCI in the lesion(s) treated with the Pan-vascular interventional robotic system, without in-hospital major adverse coronary events (MACE).
Technical Success | Procedure
  Defined as successful completion of the robotic-assisted PCI absent unplanned conversion to manual for guidewire or balloon/stent catheter inability to navigate vessel anatomy or poor guide catheter support.

SECONDARY OUTCOMES:
Procedure Time | Procedure
  Defined as the time measured from the insertion of the hemostasis sheath until the removal of the guide catheter.
PCI time | Procedure
  Defined as the time measured from the insertion of the guide catheter until the removal of the guide catheter.
Fluoroscopy Time | Procedure
  Total Fluoroscopy Time during procedure will be captured
Radiation Exposure | Procedure
  Patient and Main operator radiation exposure dose recorded by portable radiation monitor during the procedure, respectively.
Contrast agent dosage | Procedure
  The total amount of contrast agent used during the whole procedure.

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Shanghai Zhongshan Hospital, Shanghai, Shanghai Municipality
  - Kashi Prefecture Second People's Hospital, Kashgar, Xinjiang

IPD SHARING:
Plan to Share IPD: No